CLINICAL TRIAL: NCT06600139
Title: A Feasibility Study of the Collaboration-Screening-Referral Model - an Approach to Identify Parents in Child Welfare Services Who Need Mental Health Support
Brief Title: Screening to Identify Parents in Need of Mental Health Support: a Feasibility Study in Child Welfare Services
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Martin Forster, Principal Investigator, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: SSH feasibility study
Record Dates: First submitted 2024-08-23; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Mental Disorder; Depression; Anxiety; Child Abuse; Child Neglect; Child Maltreatment
Keywords: Parenting; Screening; Child Maltreatment; Depression; Anxiety
MeSH Terms: conditions — Mental Disorders; Depression; Anxiety Disorders | interventions — Models, Biological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- The Collaboration-Screening-Referral model (Experimental): The Collaboration-Screening-Referral model (in Swedish: Samverkan-Screening-Hänvisning - SSH) - an approach to screen parents involved with child welfare services for symptoms of mental illness, establish intra-agency collaboration, and facilitate referrals to mental health services. Social workers are trained to employ the SSH.
  Interventions: Behavioral: The Collaboration-Screening-Referral (SSH) model

INTERVENTIONS:
Behavioral: The Collaboration-Screening-Referral (SSH) model — The SSH aims to identify parents in need of mental health support and to strengthen social workers' competence in addressing mental illness. The SSH includes three components: 1) Collaborating - establishing collaboration with local services offering support to adults with mental illness, 2) Screening - using screening instruments for depression (the Patient Health Questionnaire - PHQ-9) and anxiety (GAD-7) to identify symptoms of mental illness among parents, and 3) Referral - Discussing the results of the screening with parents and referring to appropriate services. Techniques from motivational interviewing are included. Social workers receive training and material to administer the screening and refer parents in need of support.

SUMMARY:
The main aim of this study is to evaluate the feasibility, preliminary effects and experiences of the Collaboration-Screening-Referral approach (in Swedish: Samverkan-Screening-Hänvisning - SSH) when used with parents referred to the Swedish child welfare services. The SSH is an approach to screen parents for symptoms of mental illness using structured questionnaires, establish intra-agency collaboration, and refer to mental health services. Additionally, to increase social workers' competence in assessing and handling mental illness through receiving training in the SSH and administering the screening to parents.

The main questions the project aims to answer are:

* Are parents engaged with child welfare services willing to undergo screening for symptoms of depression and anxiety?
* How have the implementation of the SSH proceeded and to what degree is it sustained?
* How do parents and social workers experience the SSH?
* Do social workers' behaviors, knowledge and competence relevant to supporting parents with mental illness increase when implementing the SSH?

Social workers answer questions before and after their training and after 6 and 12 months. Additionally, social workers and parents will be interviewed. Qualitative and quantitative within-group analyses will be conducted to examine experiences and preliminary effects of the SSH.

DETAILED DESCRIPTION:
BACKGROUND:

Parental mental illness is prevalent and associated with several family-related risks. Parental mental illness is more common during circumstances characterized by family-related risk factors and for parents in contact with the child welfare system. Further, children to parents with mental health problems are at increased risk of developing own psychiatric problems in childhood and later adulthood. Additionally, parental mental illness influences parenting ability and is a strong risk factor for child maltreatment (CM). CM strongly increases the risk of children developing a range of psychiatric problems.

Identifying mental illness among parents within the child welfare services (CWS) and referring them to evidence-based treatment in healthcare could be essential for improving children's well-being and reducing the risk of CM. For that, intra-agency collaboration is considered crucial. Collaboration between the CWS and healthcare is however a known issue.

One way to address the lack of knowledge in assessing mental illness and support intra-agency collaboration can be routines for screening and referrals. Screening everyone in a setting can be a non-stigmatizing approach to assess symptoms and risk behaviors. Screening parents for mental health symptoms is widely implemented within pediatric healthcare, e.g., screening for post-natal depression, but is to our knowledge not a common approach within the CWS. Additionally, the lack of evidence-based methods has often been cited as a shortcoming within the CWS. Furthermore, social workers could lack the competence to identify mental illness, as it is not included in their basic education. It is therefore assumed that social workers do not always assess parents' mental health with validated procedures and do not always refer parents in need.

PURPOSE AND RESEARCH QUESTIONS:

The main aim of this project is to improve early identification of mental illness in parents reported for CM and to make treatment accessible for families with additional needs. The feasibility of the Collaboration-Screening-Referral model (in Swedish: Samverkan-Screening-Hänvisning - SSH) will be evaluated - an approach for screening parents for symptoms of mental illness and referring to support. The research questions are:

1. Are parents engaged with CWS willing to undergo screening for symptoms of depression and anxiety?
2. What barriers and facilitators to implementing the SSH have there been?
3. In what ways do parents and social workers experience that the children are influenced by the SSH, and what support the children in these families might need?
4. Do social workers' behaviors relating to assessing and handling mental illness and intra-agency collaboration procedures increase when implementing the SSH?
5. Do social workers' knowledge and perceived competence in assessing and managing mental illness increase after employing the SSH?
6. What strategies have been employed by the CWS agencies in the implementation of the SSH?
7. To what degree is usage of the SSH sustained 12 months after initiation?

METHODS:

SSH is a structured approach for screening and referring parents who need mental health support, designed for use by social workers within CWS. Municipalities will be recruited to take part in the research project and implement the SSH. First, staff will be trained in mental health screening, and a referral routine will be established. Units will also be encouraged to arrange meetings with local mental health clinics. Social workers will then administer the screening to parents. Questionnaires are followed by a discussion about well-being and support needs. The social worker can provide information on available mental health resources and offer support in establishing a contact.

The data collection will include surveys and interviews/focus groups. In connection with the training, staff will respond to a survey (baseline measurement) regarding their work methods and perceived competence in addressing mental health issues. Prior to participation, staff will be given information about the study and provide informed consent via an online platform before they access the survey. The data collection will then be divided into two phases.

Phase 1. After the first municipalities have used the SSH for approximately 3 months, social workers will participate in interviews or focus groups. If necessary, the SSH will be modified before further evaluation.

Phase 2. In the next phase, these and additional municipalities will continue to use the SSH as part of routine work. Approximately 6 months from baseline, staff will answer a follow-up survey and interviews and/or focus groups will be conducted. Further, social workers will be asked to recruit parents who have completed the screening for interviews. They will give oral information and provide a link to where parents can read written information and give informed consent. For parents who consent to participate, a person from the research team will call and inform the parent about the study, give the possibility to ask questions, and book a time for the interview. Interviews/focus groups will be conducted by phone calls or video meetings.

SAMPLE SIZE CALCULATION AND ANALYSES:

Quantitative data in surveys to staff will be presented descriptively and statistically analyzed (e.g., t-tests/non-parametric alternative). Psychometric statistics will be calculated. For a power of 80% to detect a medium sized effect (d = 0.50), the total sample size of participating staff has to be N = 34 (alpha = 0.05). To account for a drop-out rate of approximately 10%, the aim is to recruit 40 participants. Qualitative data will be analyzed employing qualitative methods, e.g., thematic analysis. For interviews, 20-40 social workers and 10-25 parents will be recruited. The specific number will be dependent upon achieving a sufficiently rich dataset according to qualitative methodological standards, e.g., data saturation or information power.

The data from the questionnaire administered to parents to assess symptoms of depression and anxiety is presented in a separate study: "Identifying Parents in Child Welfare Services Who Need Mental Health Support: Depression and Anxiety Symptoms". Based on the power calculation for that study, the aim is that 290 parents respond to the questionnaire. In this study, only the questions from parents' questionnaire assessing acceptability of the screening process are included.

ELIGIBILITY:
SOCIAL WORKERS:

Inclusion Criteria:

* Working at the participating units.

Exclusion Criteria:

* None.

PARENTS:

Inclusion Criteria:

* A parental role in relation to a child 0-17 years old (the participant does need not be a guardian or biological parent, can also be, for example, a partner to a parent).
* A child welfare report has been filed for the child or the parent has reached out to the CWS themselves.

Exclusion Criteria:

* None.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 355 (Estimated)
Dates: Start 2024-09-20 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Social workers: Change from baseline in behaviors related to assessing and assisting parents with mental health challenges | At baseline (before the training in SSH) and at 6-months follow-up
  Social workers will answer a questionnaire developed for the study, consisting of 12 questions about the methods they have used in the past months to assess and assist parents with mental health challenges. The questions are scored on a scale of 0 to 4, with a higher score indicating more frequent use of methods. Responses will be summarized to a total score of 0-48 or presented at the individual item level. Follow-up questions inquire about the specific instruments and interview guides used, the circumstances under which questionnaires are administered, and allow social workers to add additional methods in free-text.
The proportion of parents declining to complete the screening | At baseline
  Social workers will document the proportion of parents who choose not to complete the screening.

SECONDARY OUTCOMES:
Social Workers: Change from baseline in perceived competence in supporting parents with mental health challenges | At baseline and at 6-months follow-up
  A 7-item questionnaire, designed for this study, will assess social workers' perceived competence in supporting parents with mental health challenges. Each item is scored on a scale of 0 to 3, with higher scores indicating greater perceived competence. The total score ranges from 0 to 21. The results may also be presented at the individual item level.
Social workers: Description (qualitatively) of reasons not to offer the screening | At 6 months follow-up
  Social workers will provide reasons for why they have not offered the screening to parents.
Parents: Experiences of the SSH-model through individual qualitative interviews | Approximately 2-10 weeks after baseline
  Parents who have completed the screening will participate in interviews to evaluate their experiences, focusing on aspects such as acceptability and any discomfort or adverse encounters.
Social workers: Experiences of the SSH-model through interviews or focus groups | Approximately 3 and 6 months after baseline
  Social workers will participate in interviews or focus groups to evaluate their own and parents' experiences with the SSH model. The interviews will cover topics such as acceptability, the implementation process, perceived competency in assessing mental health, and the fit of the SSH with families' needs.
Social workers: Change from baseline in knowledge of mental illness | At baseline, after 2-3 weeks, and at 6-months follow-up
  Social workers will complete a knowledge test on mental illness and related methods to assess symptoms and provide support. The test includes multiple-choice questions with right or wrong answers as well as a case example where staff are asked to provide reasoning based on open-ended questions.
Social workers: Acceptability of the SSH | At 6 months follow-up
  A 4-item questionnaire, designed for the study, will be administered to social workers to assess their acceptability of the SSH. Items are scored from 0-4, with higher scores indicating greater acceptability. The responses will be summarized into a total score ranging from 0 to 16 or presented at the item level.
Parent: Acceptability of the screening | At baseline
  The questionnaire administered to parents includes three questions assessing their acceptability of the screening process. Each item is scored on a scale of 0 to 2, resulting in a total score ranging from 0 to 6, with higher scores indicating greater acceptability. Items may also be presented at the individual item level. Parents complete these questions at the end of the screening instrument.
Social workers: Experienced barriers and facilitators to parents receiving help for mental illness (qualitatively) | At 6 months follow-up
  Social workers will report perceived factors that influence whether parents receive mental health support. They will use a checklist of possible factors and provide additional details in free text.
Social workers: The number of strategies used to implement the SSH | At 6 months follow-up
  The implementation of the SSH will be assessed using a checklist completed by one social worker at each site, which will detail the implementation strategies employed.
Social workers: Experiences of the implementation of the SSH (qualitatively) | At 6 months follow-up
  A questionnaire, administered to one social worker per site, will explore potential facilitators and barriers to the implementation of the SSH through open-ended questions.
Social workers: Proportion of sites where implementation of the SSH is sustained | At 12 months follow-up
  One social worker per site will report whether they continue to utilize the SSH 12 months after implementation and provide reasons for either continuing or discontinuing its use.
Social workers: Proportion of training completion | From baseline up to 6 months follow-up
  The proportion of training completion (0% = no training, 100% = full training) will be tracked through the online platform where the training is offered and by recording attendance at live sessions.
Social workers: Background information | At baseline
  Social workers trained in the SSH will respond to questions about their background.
Parents: Background information | Approximately 2-10 weeks after baseline
  Parents who participate in interviews will be asked some questions about their background during interviews.
Social Workers: Satisfaction with online training | 1, 2 and 3 weeks from baseline
  Social workers will respond to some questions regarding satisfaction with the modules in the online training. The questions is added after each module. They are assessed on a 5-point likert scale scored from 0-4, and will be presented at the individual item level. Higher scores indicates greater satisfaction. They can also provide suggestions for improvements in free text.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Forster, PhD, Principal Investigator — Karolinska Institutet

IPD SHARING:
Plan to Share IPD: No